CLINICAL TRIAL: NCT07270120
Title: Senolytics to Improve Physical and Cognitive Function in Older Adults With Multiple Sclerosis
Brief Title: Senolytics for Secondary Progressive MS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Yinan Zhang, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20251750
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS) Secondary Progressive
Keywords: senolytic; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Dasatinib and quercetin
  Interventions: Drug: Dasatinib and quercetin

INTERVENTIONS:
Drug: Dasatinib and quercetin — Participants will receive 100 mg of dasatinib and 1250 mg of quercetin orally once a day for 2 days every 2 weeks over 12 consecutive weeks
  Other Names: D+Q

SUMMARY:
This is a clinical trial to see whether senolytic therapy is safe and feasible for patients with secondary progressive MS and whether treatment improves physical and thinking abilities. The study seeks to enroll adults with secondary progressive MS (SPMS), aged 50-85, who are not currently taking a MS disease-modifying therapy and have noticed their MS symptoms getting worse. People who join the study will take the medicines dasatinib and quercetin by mouth every two weeks for three months. These medicines work together to remove old, damaged cells that may cause inflammation and slow the repair of nerves. Participants will also be followed for one year from enrollment to monitor for treatment effects.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic immune-mediated inflammatory and neurodegenerative disorder of the central nervous system (CNS), which afflicts approximately one million people in the United States. Age is the strongest driver of disease course in MS. With increasing age, most older adults with MS develop a progressive disease phenotype characterized by gradual accrual of irreversible neurological disability, for which there are no effective treatments that reliably slow disease progression. Cellular senescence is a hallmark of aging, whereby senescent cells accumulate with age and produce mediators of inflammation through the senescence-associated secretory phenotype (SASP). In MS, senescent cells have been identified in both the central nervous system and peripheral immune compartments contributing to SASP expression, promoting chronic inflammation, axonal damage, and failure of myelin repair, and ultimately leading to functional decline. Senescent cells can be selectively removed by senolytic drugs, which delay age-related dysfunction in animal models and show potential for improving functional outcomes in human clinical trials. The senolytic drug combination of dasatinib and quercetin (D+Q) selectively induces apoptosis of senescent cells in human tissue. Our pilot data shows D+Q treatment improves function and survival in experimental autoimmune encephalomyelitis, the widely used animal model of MS. Emerging evidence from early phase clinical trials of D+Q in age-related diseases shows improvement of gait speed in idiopathic pulmonary fibrosis and CNS penetrance of dasatinib in Alzheimer's disease. However, studies of senolytic therapy for people with MS have yet to be conducted. The investigators hypothesize that treatment with D+Q will be well tolerated, improve physical and cognitive function, reduce circulating biomarkers of senescence and neurodegeneration, and attenuate T-cell immune exhaustion. The investigators will test this hypothesis through a single arm, open label, study to 1) determine the feasibility of 3 months of intermittent D+Q treatment in 30 older adults age 50-85 with secondary progressive MS and 2) to obtain preliminary data of D+Q treatment on physical and cognitive function and 3) serum biomarkers of senescence, neurodegeneration, and the circulatory T cell repertoire. Targeting cellular senescence represents a novel strategy for treating progressive MS, and results from the study will lay the foundation for a future randomized controlled trial of senolytics to treat progressive MS.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 50-85 with SPMS diagnosed using the 2024 McDonald Criteria
2. Not treated with a DMT for MS within the last 6 months or have used alemtuzumab, cladribine, or mitoxantrone.
3. Evidence of MS progression over the past 12 months.

Exclusion Criteria:

1. Unstable coronary artery disease (myocardial infarction within 6 months or angina)
2. Hospitalization within 6 months
3. Stroke or transient ischemic attack in the past 6 months
4. Pulmonary arterial hypertension
5. Current or chronic history of liver disease
6. Alzheimer's or Parkinson's disease
7. Drug or alcohol abuse in the previous 5 years
8. History of coagulation disorders, central nervous system hemorrhage, or gastrointestinal hemorrhage
9. History of angina or myocardial infarction, arrhythmia, or heart failure at any time
10. QTc prolongation
11. Anemia (Hgb<9), thrombocytopenia (platelets<50,000 per microliter), or neutropenia (ANC< 1000 per microliter)
12. Moderate hypokalemia (2.9 mmol/L) and moderate hypomagnesemia (0.9-1.1 mg/dL or 0.37-0.45 mmol/L)
13. ALT/AST >1.5x ULN, total bilirubin >ULN, and alkaline phosphatase >2x ULN
14. Chronic renal disease (glomerular filtration rate < 30 mL/min/1.73 m2)
15. Alcohol intake greater than 2 drinks/day for men and greater than 1 drink/day for women
16. Anti-arrhythmic medications known to cause QTc prolongation
17. Antipsychotics and anxiolytics
18. Anti-platelet or anti-coagulant medications other than aspirin
19. Quinolone antibiotics
20. Pregnant or lactating subjects or subjects intending to become pregnant or to donate egg/sperm
21. Participants with p16INK4a below the median of SPMS patients in the OSU Aging and MS Cohort
22. Use of drugs metabolized by the same liver enzymes as D or Q

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Participant retention rate | Baseline until 3 months
  Participant retention rate with D+Q therapy with no more than one missed study visit
Recruitment feasibility | Baseline
  The number of subjects screened to identify eligible participants
Frequency of adverse drug effects of dasatinib and quercetin | From baseline through study completion at 1 year
  Frequency of adverse drug effects of dasatinib and quercetin

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State Martha Morehouse Outpatient Care, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data management and sharing plan will be consistent with the NIH Data Sharing Policy and Implementation Guidance which recognizes the need to make the research data generated from the NIH support projects available to the scientific community while ensuring that the privacy and autonomy of research participants are respected, and that confidential/proprietary data are appropriately protected. Data will include demographic, clinical, functional, and cognitive data from study participants, in addition to banked blood, urine, and lymphocytes. All investigators wishing to access the data will submit a brief proposal to Drs. Zhang or Kirkland describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Dr. Zhang and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working electronic data file and appropriate documentation.